CLINICAL TRIAL: NCT00873353
Title: An Open Non-randomized Multicenter Phase II Trial to Evaluate the Efficacy and Safety of Tarceva in Combination With Capecitabine in Patients With Advanced Pancreatic Cancer
Brief Title: Trial to Evaluate the Efficacy and Safety of Tarceva and Capecitabine in Advanced Pancreatic Cancer Patients
Acronym: XELTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Gallego de Investigaciones Oncologicas (Other)
Responsible Party: Rafael López López, Grupo Gallego de Investigaciones Oncologicas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21154; 2007-003206-96 (EudraCT Number)
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2010-08

CONDITIONS: Metastatic Adenocarcinoma of the Pancreas
Keywords: Metastatic Adenocarcinoma of the Pancreas
MeSH Terms: interventions — Capecitabine; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Unique arm (Experimental): 6 cycles (3 weeks each one) of :
  * capecitabine 1000mg/m2, bid, oral. Days: 1-14 every three weeks
  * erlotinib (Tarceva®) 150mg/day, oral. Days: every days
  Interventions: Drug: capecitabine + erlotinib

INTERVENTIONS:
Drug: capecitabine + erlotinib — 6 cycles (3 weeks each one) of :
  * capecitabine 1000mg/m2, bid, oral. Days: 1-14 every three weeks
  * erlotinib (Tarceva®) 150mg/day, oral. Days: every days
  Other Names: capecitabine (Xeloda®)y erlotinib (Tarceva®)

SUMMARY:
The purpose of this study is to determine efficacy of the treatment with erlotinib in combination with capecitabine in patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
This efficacy will be determined by objective response rate following RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent
2. Informed consent signed by the patient
3. Age > 18 years old
4. Able to fulfill all criteria from the protocol
5. Performance status Karnofsky ≥ 60% (ECOG 0-2)
6. Life expectancy ≥ 12 weeks
7. Histologically or cytological (excluding endocrine pancreatic tumour), with metastatic (stage IV), following 6th edition of TNM classification
8. Measurable disease following RECIST criteria
9. Adequate bone marrow function as determined by:

   * Absolute Neutrophil account (ANC) ≥ 1,5 x 109/L
   * Platelets: ≥ 100 x 109/L
   * Hemoglobin: ≥ 9 g/dL.
10. Adequate liver function, as determined by:

    * Serum bilirubin (total): ≤ 1,5 x LSN
    * AST, ALT ≤ 2,5 x LSN in patients without liver metastasis. In patients with liver metastasis ≤ 5 x LSN
11. Adequate renal function, as determined by:

    * Clearance creatinine > 60.0 ml/min
12. Men or women potentially fertile (including postmenopausal women amenorrheic at least 24 months before the study) should use adequate contraceptive methods (oral contraceptives, intrauterine disposal, barrier methods together with spermicide or surgery sterilization)

Exclusion Criteria:

1. Local pancreatic cancer (stage IA-IIB) or locally advance cancer (stage III), following the TNM 6th edition classification. Patients with metastatic disease that relapse after the initial diagnosis of local or advance disease could be included in this study.
2. Evidence of medullary compression, carcinomatosis meningitis or brain metastasis. In case of clinical suspicious of brain metastasis is mandatory to perform a brain TAC/MR 4 weeks prior inclusion.
3. Previous systemic treatment for metastasis pancreas cancer. Adjuvant chemotherapy is permitted ≥ 4 weeks prior de inclusion. All toxicities from the adjuvant treatment must been solve before the inclusion and should be confirmed the diseases progression (metastatic disease) alter adjuvant treatment
4. Primary tumours Developer 5 years previous to the inclusion, except in situ cérvix carcinoma or skin basocellular cancer properly treated
5. Non-controlled hypertension or cardiovascular disease clinically significant (active):

   * Cerebrovascular accident/ictus (≤ 6 weeks prior to inclusion)
   * Heart attack (≤ 6 months prior to inclusion)
   * Instable angina
   * Congestive cardiac insufficiency (grade II or superior following to New York Heart Association (NYHA)
   * Severe cardiac arrhythmia that require medication
6. Significant ophthalmology anomalies
7. Deficit in dihydropyrimidine dehydrogenase (DPD)
8. Unable to take oral drug. Previous surgical process that affect the absorption or make the needed to have intravenous feeding or parenteral nutrition with lipids.
9. Pregnancy women or in latency period. Negative pregnancy test needed 7 days prior to initiation drug study
10. Actual or 30 days previous to study treatment with other investigational drug or participation in other trial
11. Previous treatment with Capecitabine or EGFR inhibitor.
12. Any other disease, metabolic disease
13. Known hypersensibility to any study drug or any of their component, or to 5-fluorouracile

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Objective response rate following RECIST criteria | within study period

SECONDARY OUTCOMES:
Overall survival | within study period
6 months survival rate | within first 6 months after study inclusion
Progression Free Survival (PFS) | Time from study inclusion to disease progression
Time to treatment failure (TTF) | Time from study inclusion to treatment failure
To determine the index of clinical benefit | at the end of the study
To determine the safety and tolerability of erlotinib and capecitabine when administered together | Within study period

CONTACTS AND LOCATIONS:
Overall Officials: Rafel López López, Coordinator, Study Chair — Grupo Gallego de Investigaciones Oncológicas
Locations (8):
- Spain (8):
  - Complejo Hospitalario Universitario de La Coruña, A Coruña, La Coruña
  - Centro Oncológico de Galicia, A Coruña, La Coruña
  - Hospital Arquitecto Marcide, Ferrol, La Coruña
  - Complejo Hospitalario Xeral Calde, Lugo, Lugo
  - Complejo Hospitalario de Orense, Ourense, Orense
  - Hospital do Meixoeiro, Vigo, Vigo
  - Complejo Hospitalario Xeral Cies, Vigo, Vigo
  - Hospital POVISA, Vigo, Vigo